CLINICAL TRIAL: NCT04132700
Title: Longitudinal Evaluation of Energy Expenditure in ICU Patients From Admission to Discharge Using A Novel Indirect Calorimeter: LEEP-Forward Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: LEEP-COVID study (NCT04350073) initiation enables inclusion of COVID-positive subjects
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00103738
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2019-11

CONDITIONS: Metabolism Requirement; Energy Requirement; Indirect Calorimetry
Keywords: energy expenditure; respiratory quotient; Intensive Care Unit (ICU); indirect calorimetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ICU Patients (Experimental): Patients admitted to the ICU will be monitored using the Q-NRG for up to 30 mins.
  Interventions: Device: Q-NRG Metobolic Cart Device

INTERVENTIONS:
Device: Q-NRG Metobolic Cart Device — ICU pateints will be measured using the Q-NRG device for up to 30 mins. These measurements will take place every other day while the patients are in the ICU. Then they will occur a minimum of 3 times a week until discharge.

SUMMARY:
The purpose of this study is to utilize the new indirect calorimetry Q-NRG device to the measurement of energy expenditure (EE) throughout your intensive care unit (ICU) stay and ultimately address fundamental questions about metabolism and energy requirements for critically ill patients. The study will use a new, investigational calorimeter called the Q-NRG (the study device, supplied by Cosmed, Italy). The word "investigational" means the study drug or device or biologic is still being tested in research studies and is not approved by the U.S. Food and Drug Administration (FDA). A calorimeter is a device that connects to your breathing machine tubing for a short period (about 30 minutes) and helps to determine what nutrition you may need in your current condition.

There are FDA approved calorimeters that have been used as the current standard of care. These devices and the new Q-NRG calorimeter measure oxygen consumption and carbon dioxide production (the gas you breathe out when you exhale) and calculate energy expenditure. Unfortunately, previously existing calorimeters are complicated to use, cumbersome and require time for measurements. It is hoped the new calorimeter will be easier and more practical to use and, through the measurements we take, we will have a better understanding of a patient's caloric needs for healing.

Muscle mass and quality play a role in determining EE and metabolic needs. Massive loss of muscle mass and quality that occurs in critical illness significantly affects EE and nutritional needs and should be accounted for in clinical nutrition delivery. Imaging (standard of care abdominal CT and MSK ultrasound) will be used to assess muscle mass, and muscle quality (amount of intramuscular adipose content; IMAT).

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients requiring mechanical ventilation for > 48 hours
* Patients admitted to Duke Surgical/Trauma ICU, Medical ICU, Cardiothoracic ICU, and Neuro ICU
* Patients must be enrolled within 72 hours of ICU admission

Exclusion Criteria:

* Fraction of inhaled oxygen (FIO2) > 70%
* Positive end expiratory pressure (PEEP) > 10cmH2O
* Peak ventilatory pressure > 30cmH20
* Presence of air leaks from thoracic drain tube
* Changes in vasoactive agent dose (>20%, <1 hr before or during IC)
* Agitation or change in sedative/analgesic dose (>20%, <1 hr before and/or during IC)
* Change in body temperature (>0.5°C, <1 hr before and/or during IC)
* Expected duration of ICU stay < 24 hours
* Expected survival of the patient < 24 hours
* Continuous Renal Replacement Therapy (CRRT/CVVH that does not experience an appropriate interruption of at least 60 minutes to allow for indirect calorimetry measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Resting Energy expenditure(REE) over time, as measured by the indirect calorimetry Q-NRG device | Minimum of every other day while in ICU (up to 10 days). Once discharged from ICU minimum of 3x a week until discharge (up to 3 weeks)
  The amount of CO2 produced combined with O2 consumed is called the REE (kcal/day) and is measured by the gases exchanged at the mouth.
Changes of the Respiratory Exchange Ratio (RER) as measured by the indirect calorimetry Q-NRG device | Minimum of every other day while in ICU (up to 10 days). Once discharged from ICU minimum of 3x a week until discharge (up to 3 weeks)
  RER (ratio of CO2 produced to O2 consumed is called the respiratory exchange ratio (RER) and is measured by the gases exchanged at the mouth

SECONDARY OUTCOMES:
Changes of Intramuscular adipose tissue (IMAT) content from the psoas at the Level of L3/Th3 | Minimum of every other day while in ICU (up to 10 days). Once discharged from ICU minimum of 3x a week until discharge (up to 3 weeks)
  the change over time of CT-derived area of intramuscular adipose tissue in cm2
Changes of Intramuscular adipose tissue (IMAT) from rectus femurs - vastus laterals - temporalis - styloglossys | Minimum of every other day while in ICU (up to 10 days). Once discharged from ICU minimum of 3x a week until discharge (up to 3 weeks)
  the change over time of Ultrasound-derived area of intramuscular adipose tissue in %

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wischmeyer, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No